CLINICAL TRIAL: NCT04330170
Title: Inferior Vena Cava Filters Utilization in Patients With Venous Thromboembolism: Analysis of a Database of a Tertiary Hospital
Brief Title: Inferior Vena Cava Filters: Analysis of a Database
Status: Completed | Type: Observational
Sponsor: Pirogov Russian National Research Medical University (Other)
Responsible Party: Principal Investigator, Igor Zolotukhin, Professor of Surgery, Pirogov RNRMU, Zolotukhin Igor Anatolievich, Pirogov Russian National Research Medical University
Other Study IDs: 180
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Deep Vein Thrombosis, Pulmonary Embolus
Keywords: deep vein thrombosis; inferior vena cava-filter; pulmonary embolism
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study a retrospective analysis of patients database was performed, who underwent treatment for deep vein thrombosis in tertiary hospital by using inferior vena cava-filters

DETAILED DESCRIPTION:
The aim of this research was to assess the cava-filter implantation frequency in a tertiary hospital with venous thromboembolism treatment center.

A retrospective analysis of patient's database was performed, who underwent treatment in the tertiary clinic between 2016 - 2017. In total, 2399 patients with venous thromboembolism were hospitalized, 442 cava-filters were implanted (239 in 2016 and 203 in 2017), which accounted for 18.4% of patients with venous thromboembolism. Removable cava-filters models were used in most cases (98.8%). Contraindications for anticoagulation were reason for cava-filters implantation in 119 (26.9%) cases, and in 184 patients (41.6%) cava-filters were implanted due to the inefficiency of anticoagulation. 38 (8.6%) patients with deep vein thrombosis (DVT) and pulmonary embolism had pulmonary hypertension of the 2nd to 3rd degree, which caused the implantation of cava-filters .

The occlusion of the inferior vena cava and cava-filters verified in 116 (26.9%) patients after cava-filters implantation, based on repeated ultrasound. The overall mortality rate in the group of patients with venous thromboembolism was 0.25% (6 patients), 5 of them (1.1%) underwent cava-filters implantation. The cause of all lethal outcomes was the progression of the underlying disease. During the next hospitalization 29 (6.5%) of implanted filters were endovascularly removed.

There are 18.4% of patients with venous thromboembolism undergoing cava-filters implantation for various reasons in a tertiary hospital. At the same time, occlusion of the inferior vena cava and cava-filters in the early post implantation period is observed in 26.9%. However, without clear criteria for the differentiation of cava-filters embolism from its thrombosis, we cannot assess whether this was a complication, or if the cava-filters completed its task by preventing pulmonary embolism. Thus, the validity of implanting cava filters question in terms of efficiency and safety remains unanswered, which poses the task for deep study of this problem and thorough analysis of the indications for the cava-filters implantation.

ELIGIBILITY:
Inclusion Criteria:

* Anticoagulation therapy contraindicated
* Anticoagulation therapy ineffective
* High pulmonary embolism risk (floating thrombus in proximal location)
* Deep vein thrombosis/pulmonary embolism together with high pulmonary hypertension(>50 mm.Hg)

Ages: 16 Years to 91 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 2399 patients who were either hospitalized with venous thromboembolism or diagnosed with venous thromboembolism during hospital stay in 2016-2017. Of them there were 1173 male (48,9%) and 1226 female (51,1%) patients with average age of 62,4 ± 15,2 (min - 16, max - 96).
Sampling Method: Probability Sample
Enrollment: 2399 (Actual)
Dates: Start 2016-01-13 (Actual); Primary Completion 2020-03-28 (Actual); Study Completion 2020-03-28 (Actual)

PRIMARY OUTCOMES:
Number of participants with occlusion of inferior vena cava-filter | from date of inferior vena cava-filter implantation until the date of discharge, up to 1-2 weeks
  Number of participants with embolic or thrombotic occlusion of inferior vena cava-filter

SECONDARY OUTCOMES:
Number of participants who have undergone cava-filter removal | from date of inferior vena cava-filter implantation until the date of discharge, up to 1-2 weeks
  Number of participants , who underwent retrieving of cava-filter due to the pulmonary embolism risk regression
Number of participants with implanted cava filter in whom the filter remained intact | from date of inferior vena cava-filter implantation until the date of discharge, up to 1-2 weeks
  Number of participants with filter implanted without the possibility of its removal due to various reasons and without its occlusion

CONTACTS AND LOCATIONS:
Locations (1):
- The Federal Budget-Funded Institution National Medical Surgical Center named after N. I. Pirogov of the Ministry of health of the Russian Federation, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No